CLINICAL TRIAL: NCT01757509
Title: A Randomized Controlled Feasibility Trial to Determine the Effectiveness of Set Dancing for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Joanne Shanahan, Joanne Shanahan, B.S.c, MISCP, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST1
Record Dates: First submitted 2012-12-01; First posted 2012-12-31 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Set dancing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Other): Participants in this group will receive a set dancing intervention along with their usual care.
  Interventions: Other: Intervention group
- Control Group (No Intervention): The control group will continue with their usual medical regime, activities of daily living and exercise habits and at the end of the study participants in this group will be offered the set dancing intervention.

INTERVENTIONS:
Other: Intervention group — Participants will attend eight weeks of set dancing classes. Each class will be one and a half hours. Family members or volunteers will partner each participant with Parkinson's disease. The class will be led by a Chartered Physiotherapist who is also a set dancing teacher. Set dancing steps and sets will be thought and progressed in line with the participants' abilities. Frequent rests will be taken during the class.
  Participants will be given a home exercise programme which will involve mental rehearsal, listening to music, watching dance DVD's and practicing dance material in the seated position to reduce the risk of falling.
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate if set dancing is beneficial and feasible for those with Parkinson's disease in Ireland. The hypothesis of this feasibility study are that:

* Participants will be able to partake fully in the intervention without reporting adverse events.
* There will be evidence of gains in functional exercise tolerance, balance, motor performance and quality of life in those with Parkinson's disease who participate in eight weeks of set dancing classes compared to a control group.

DETAILED DESCRIPTION:
Background: Previous research has found that people with Parkinson's disease who participate in dance classes have improved functional exercise capacity, mobility, balance and quality of life (Duncan and Earhart 2012; Hackney and Earhart 2009). Dance may be an effective intervention for people with Parkinson's disease as it targets key components of rehabilitation programmes for people with Parkinson's disease (Earhart 2009). These components include use of cueing strategies, training of muscle power and balance and focusing of attention on movement strategies.

The benefit of many forms of dance have being investigated in people with Parkinson's disease including Tango, (Hackney et al 2007), Contact Improvisation (Marchant et al 2010) and modern dance (Batson 2010). However, recently Irish set dancing has also being found to be beneficial for those with Parkinson's disease (Volpe et al 2013). Irish Set dancing may be beneficial for people with Parkinson's disease as it involves continuous movement initiation and cessation along with focusing of attention on body posture and foot placement. However, research to date has not been conducted in the Irish population. It is important to investigate if set dancing is beneficial for people with Parkinson's disease in Ireland as results may be influenced by the familiarity which the Irish population has for set dancing.

The objectives of the study are:

* To compare functional exercise tolerance, balance, motor performance and quality of life in those with Parkinson's disease before and after participating in set dancing classes, using the following validated outcome measures: Unified Parkinson's Disease Rating Scale 3, Berg Balance Scale, The Parkinson's Disease Questionnaire and The Six-Minute Walk Test.
* To compare functional exercise tolerance, balance, motor performance and quality of life in those with Parkinson's disease participating in set dancing classes to those receiving usual care.
* To assess the effect of the intervention on care giver burden using the Zarit Care Giver Burden Interview.

Participants, who meet inclusion/exclusion criteria, will be randomly assigned to a group who will receive a set dancing intervention along with their usual care or to a control group who will continue with their usual care only. Participants will be assessed the week before the intervention period begins and the week after the intervention period ends using valid and reliable outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of idiopathic Parkinson's disease (Hackney et al 2007; Marchant et al 2010), stage 1-2.5 on the Hoeln and Yahr scale for staging of Parkinson's disease (Batson 2010)
* Showing a clear benefit from anti-Parkinson medication (Marchant et al 2010)
* Able to walk three meters with or without an assistive device (Hackney and Earhart 2009)
* Not pregnant
* Over 18 year of age
* Have a TV and DVD player in their own home to allow them to participate in the home exercise programme.

Exclusion Criteria:

* A serious cardiovascular and/or pulmonary condition (Lodder et al 2004)
* A neurological deficit other than Parkinson's disease (Batson 2010; Marchant et al 2010)
* Evidence of a musculoskeletal problem contraindicating participation in exercise participation(Duncan and Earhart 2012)
* A cognitive or hearing problem which will effect their ability to follow instructions or hear the music (Batson 2010)
* Participated in regular dance classes in the past six months (Marchant et al 2010)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (To assess change in balance) | This outcome will be assessed the week before the intervention begins and the week after the intervention period ends.
  The aim of the Berg Balance Scale is to assess functional balance (Marigold and Eng 2006). The measure consists of 14 items. Each item requires the participant to perform a functional balance task such as turning, stepping and reaching (Marigold and Eng 2006). A lower score is indicative of compromised balance performance. This measure is a valid and reliable measure and has being found to correlate with UPDRS scores and Hoeln and Yahr scale for staging of Parkinson's disease (Qutubuddin et al 2005).

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale 3 (UPDRS-3) (To assess changes in motor impairment) | This outcome will be assessed the week before the intervention begins and the week after the intervention period ends.
  UPDRS-3 is a motor subscale of the UPDRS. It is a measure of disease severity (Hackney et al 2007). The motor subscale examines various motor impairments which are associated with Parkinson's disease such as speech, tremor at rest, rigidity and gait (Heiberger et al 2011). Higher scores indicate more severe disease stage. This is a disease specific measure which is valid (Hackney et al 2007) and reliable with an excellent Intra-Class Correlation Co-efficient for test re-test reliability (Siderowf et al 2002), and intra-rater reliability (Metman et al 2004).
The Parkinson's Disease Questionnaire (PDQ-39) (To assess change in health related quality of life) | This outcome will be assessed the week before the intervention begins and the week after the intervention period ends.
  PDQ-39 will be used to assess health related quality of life (Marchant et al 2010). This questionnaire assesses the impact of Parkinson's disease in eight different areas including mobility, emotional well-being and communication. It has being found to be the most appropriate outcome measure to assess the impact of Parkinson's disease on health related quality of life as it is a disease specific test that is valid and reliable (Hackney et al 2009). Previous research has also found that this measure can detect changes in health related quality of life in response to physical activity interventions (Jenkinson et al 1997).
Six-Minute Walk Test (To assess change of functional exercise tolerance) | This outcome will be assessed the week before the intervention begins and the week after the intervention period ends.
  The six-minute walk test will be used to asses functional exercise tolerance (Falvo and Earhart 2009). This test requires participants to walk along a pre measured pathway for six minutes. This test is valid, reliable (Demers et al 2001; Schenkman et al 1997) and clinically applicable as it is simple to reproduce and reflects endurance needed for activities of daily living (Enright 2003). In previous studies, this test has detected changes in exercise tolerance in those with Parkinson's disease who completed a dance intervention (Hackney and Earhart 2009).
Zarit Care Giver Burden Interview (ZCBI)(To assess changes in caregiver burden) | This outcome will be assessed the week before the intervention begins and the week after the intervention period ends.
  ZCBI provides a multidimensional assessment of caregiver burden (Ankri et al 2005). The aim of this measure is to assess changes in caregiver burden over time (Hackney et al 2010). It consists of 22 items. Higher scores indicate greater caregiver burden (Hackney et al 2010). It is a valid and reliable measure for assessing the burden of caregivers involved in caring for those with Parkinson's disease (Martínez-Martín et al 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Meg E Morris, Prof., Study Chair — Department of Physiotherapy, School of Allied Health, La Trobe University, Bundoora 3086, Australia
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

REFERENCES:
- [Background] Hackney ME, Earhart GM. Effects of dance on gait and balance in Parkinson's disease: a comparison of partnered and nonpartnered dance movement. Neurorehabil Neural Repair. 2010 May;24(4):384-92. doi: 10.1177/1545968309353329. Epub 2009 Dec 14. PMID 20008820
- [Background] Hackney ME, Kantorovich S, Levin R, Earhart GM. Effects of tango on functional mobility in Parkinson's disease: a preliminary study. J Neurol Phys Ther. 2007 Dec;31(4):173-9. doi: 10.1097/NPT.0b013e31815ce78b. PMID 18172414
- [Background] Marchant D, Sylvester JL, Earhart GM. Effects of a short duration, high dose contact improvisation dance workshop on Parkinson disease: a pilot study. Complement Ther Med. 2010 Oct;18(5):184-90. doi: 10.1016/j.ctim.2010.07.004. Epub 2010 Aug 21. PMID 21056841
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886